CLINICAL TRIAL: NCT05420493
Title: This is a Phase I Clinical Study to Evaluate the Safety and Efficacy of CAR-T Infusion Preparation in the Treatment of CD19-positive Relapsed/Refractory Non-Hodgkin Lymphoma.
Brief Title: Clinical Study of Chimeric Antigen Receptor T Lymphocytes (CAR-T) in the Treatment of Relapsed/Refractory Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC033
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-11

CONDITIONS: Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Non Hodgkin Lymphoma
Keywords: CAR-T
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous of CAR-T (Experimental): Infusion of CAR-T cells by dose of 3-10 x105 cells/kg
  Interventions: Biological: CAR-T cells

INTERVENTIONS:
Biological: CAR-T cells — Drug: CAR-T cells； Administration method: intravenous infusion； Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion.

SUMMARY:
This is a phase I clinical study to evaluate the safety and efficacy of CAR-T infusion preparation in the treatment of CD19-positive relapsed/refractory non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label study. After meeting the eligibility criteria and enrolling on the trial, patients will undergo leukapheresis for collection of autologous lymphocytes. Once cells have been manufactured, patients will then proceed to lymphodepleting chemotherapy with cyclophosphamide and fludarabine for 1-2 consecutive days followed by the infusion of CAR T-cells at a target dose of 3-10x105 cells/kg.

ELIGIBILITY:
Inclusion Criteria:

1. CD19-positive non-Hodgkin lymphoma confirmed by cytology or histology according to WHO2016 criteria:

   1. Diffuse large B-cell lymphoma: including unspecified (DLBCL, NOS), chronic inflammation-related DLBCL, primary cutaneous DLBCL (leg type), EBV-positive DLBCL (NOS); and high-grade B-cell lymphoma (including high-grade B-cell lymphoma, NOS, and high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements); and primary mediastinal large B-cell lymphoma; and T-cell-rich histiocytosis B-cell lymphoma; and transformed DLBCL (such as follicular lymphoma, chronic lymphocytic leukemia/small B-lymphocytic lymphoma transformed DLBCL); patients with the above tumor types have been treated with at least first- and second-line drugs and have stable disease for ≤12 months , or when the best Disease progression after efficacy; or disease progression or relapse after autologous stem cell transplantation ≤12 months;
   2. According to WHO2016 criteria cytology or histology confirmed CD19 positive: follicular cell lymphoma. Patients with this tumor type have received at least third-line therapy, and recurrence or disease progression has occurred within 2 years after third-line therapy or more. Currently in disease progression, stable disease, or partial remission;
   3. According to WHO2016 standard cytology or histology confirmed CD19 positive: mantle cell lymphoma. Such patients have not been cured or relapsed after at least three-line treatment and are not suitable for stem cell transplantation or relapse after stem cell transplantation;
2. Age ≥18 years old (including the threshold);
3. According to the 2014 version of Lugano criteria, there is at least one two-dimensional measurable lesion as the evaluation basis: for intranodal lesions, it is defined as: long diameter >1.5cm; for extranodal lesions, long diameter should be >1.0cm;
4. Eastern Cooperative Oncology Group activity status score ECOG score 0-2;
5. The venous access required for collection can be established, and there are enough cells collected by non-mobilized apheresis for CAR-T cell production;
6. Liver and kidney function, cardiopulmonary function meet the following requirements:

   * Serum creatinine≤2.0×ULN;
   * Left ventricular ejection fraction ≥ 50% and no obvious pericardial effusion, no abnormal ECG;
   * Blood oxygen saturation ≥92% in non-oxygen state;
   * Blood total bilirubin≤2.0×ULN (except without clinical significance);
   * ALT and AST≤3.0×ULN (with liver tumor infiltration≤5.0×ULN);
7. Be able to understand and voluntarily sign the informed consent.

Exclusion Criteria:

1. Received CAR-T therapy or other gene-modified cell therapy before screening;
2. Received anti-tumor therapy (except systemic immune checkpoint inhibition or stimulation therapy) within 2 weeks or 5 half-lives (whichever is shorter) before screening. 3 half-lives are required to enroll (eg, ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 receptor agonist, 4-1BB receptor agonist, etc.);
3. Those who have received hematopoietic stem cell transplantation (ASCT) within 12 weeks before apheresis, or who have previously received allogeneic hematopoietic stem cell transplantation (HSCT), or those who have solid organ transplantation; immunosuppression is required within 2 weeks before apheresis Grade 2 and above GVHD of the drug;
4. Patients with atrial or ventricular lymphoma involvement or need urgent treatment due to tumor mass such as intestinal obstruction or vascular compression;
5. Have been vaccinated with live attenuated vaccine within 6 weeks before clearing the leprosy;
6. Cerebrovascular accident or epilepsy occurred within 6 months before signing the ICF;
7. History of myocardial infarction, cardiac bypass or stent, unstable angina or other clinically significant heart disease within 12 months prior to signing the ICF;
8. Active or uncontrolled autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus), except those that do not require systemic treatment;
9. Malignant tumors other than non-Hodgkin lymphoma within 5 years prior to screening, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, Ductal carcinoma in situ;
10. Uncontrollable infection within 1 week before screening;
11. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is greater than the normal reference range; or hepatitis C virus (HCV) antibody positive and peripheral blood C Hepatitis virus (HCV) RNA titer test is greater than the normal reference range; or human immunodeficiency virus (HIV) antibody positive; or syphilis test positive; cytomegalovirus (CMV) DNA test positive;
12. Women who are pregnant or breastfeeding; or women of childbearing age who have a positive pregnancy test during the screening period; or male or female patients who are unwilling to use contraception from the time of signing the informed consent form to 1 year after receiving CAR-T cell infusion;
13. Other investigators deem it inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after CAR-T cells infusion [Safety and Tolerability] | 28 days
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
Objective response rate after CAR-T cells infusion [Effectiveness] | 3 months
  Objective response rate includes CR,PR

SECONDARY OUTCOMES:
AUCS of CAR-T cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
CMAX of pCAR-19B cells [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of pCAR-19B cells expanded in peripheral blood
TMAX of pCAR-19B cells [Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of pCAR-19B cells[Cell dynamics] | 3 months
  IL-6 levels measured by Chemiluminescence method

OTHER OUTCOMES:
Objective response rate (ORR) of CAR-T treatment in patients with Relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 2 years
  Objective response rate includes：CR、PR
Overall survival(OS)of CAR-T treatment in patients with Relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 2 years
  OS will be assessed from the first CAR-T cell infusion to death from any cause
Progress-free survival(PFS) of CAR-T treatment in patients with Relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 2 years
  PFS will be assessed from the first CAR-T cell infusion to death from any cause or the first assessment of progression
Duration of Response (DOR) of CAR-T treatment in patients with Relapsed/refractory B-cell non-Hodgkin lymphoma[Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/PR to the first assessment of recurrence or progression of the disease or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Bi, M.D, Principal Investigator — Shandong Second Provincial General Hospital
Locations (1):
- Shandong Second Provincial General Hospital, Jinan, Shandong, China